CLINICAL TRIAL: NCT05684289
Title: A Phase 1, 2-Part, Randomized, Double-Blind, Placebo-controlled, Multiple Dose Study to Test the Potential Interaction of a PDE5 Inhibitor With BMS-986278 and to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986278 in Healthy Adult Participants (Part 1) and in Japanese Participants (Part 2)
Brief Title: A Study Investigating the Safety, Tolerability, Drug Levels and Drug Effect of BMS-986278 in Healthy Adult Participants (Part 1) and Japanese Participants (Part 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM027-1017
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants
Keywords: BMS-986278; Idiopathic Pulmonary Fibrosis (IPF); Sildenafil
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: BMS-986278 + Sildenafil (Experimental)
  Interventions: Drug: BMS-986278; Drug: Sildenafil
- Part 1: Placebo + Sildenafil (Placebo Comparator)
  Interventions: Drug: Sildenafil; Drug: Placebo
- Part 2: BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
  Arms: Part 1: BMS-986278 + Sildenafil; Part 2: BMS-986278
Drug: Sildenafil — Specified dose on specified days
  Arms: Part 1: BMS-986278 + Sildenafil; Part 1: Placebo + Sildenafil
Drug: Placebo — Specified dose on specified days
  Arms: Part 1: Placebo + Sildenafil; Part 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels and drug effect of BMS-986278 in healthy adult participants and Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the Japanese cohort (Part 2) must be first generation Japanese (born in Japan, not living outside of Japan > 10 years, both parents ethnically Japanese).
* Body mass index (BMI) of 18.0 kilogram (kg)/meter (m)^2 through 32.0 kg/m^2, inclusive. BMI = weight (kg)/(height [m])^2.
* Body weight ≥ 50 kg for males and ≥ 45 kg for females.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any gastrointestinal (GI) disease or surgery (including cholecystectomy) or other procedures (for example, bariatric procedures) that could affect drug absorption, distribution, metabolism, and excretion.
* Any major surgery within 4 weeks of first study intervention administration.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Mean placebo-corrected change from baseline in systolic blood pressure (SBP) (Part 1) | Up to 16 days
Maximum observed plasma concentration (Cmax) (Part 2) | Up to 14 days
Time of maximum observed plasma concentration (Tmax) (Part 2) | Up to 14 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) (Part 2) | Up to 14 days

SECONDARY OUTCOMES:
Cmax (Part 1 and 2) | Up to 16 days
Tmax (Part 1) | Up to 16 days
AUC(0-T) (Part 1) | Up to 16 days
Number of participants with adverse events (AEs) (Part 1 and 2) | 30 days after last dose
Number of participants with serious adverse events (SAEs) (Part 1 and 2) | 30 days after last dose
Number of participants with clinical laboratory abnormalities (Part 1 and 2) | 30 days after last dose
Number of participants with physical examination abnormalities (Part 1 and 2) | 30 days after last dose
Number of participants with vital sign abnormalities (Part 1 and 2) | 30 days after last dose
Number of participants with electrocardiogram (ECG) abnormalities (Part 1 and 2) | 30 days after last dose
Mean placebo-corrected change in diastolic blood pressure (DBP) (Part 1) | 30 days after last dose
Area under the concentration-time curve in 1 dosing interval (AUC [TAU]) (Part 2) | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - Syneos Health Clinical Research Services, Llc, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html